CLINICAL TRIAL: NCT05030727
Title: Comprehensive Assessments of Intraoperative NGAL Level in Geriatric Patients Undergoing Laparotomy'
Brief Title: Intraoperative NGAL Level in Geriatric Patients Undergoing Laparotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Meliha Orhon, assistant professor, Marmara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09.2021.392
Record Dates: First submitted 2021-06-04; First posted 2021-09-01 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Geriatric Presentation of Urinary Tract Infection; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of intraoperative NGAL levels in terms of acute kidney injury in geriatric patients (Other): only one group
  Interventions: Diagnostic Test: record of pNGAL

INTERVENTIONS:
Diagnostic Test: record of pNGAL — Preoperative (0.hour baseline), postoperative 24.,48. BUN, Creatinine, Lactate values in the blood of the patients at 1 hour, and for plasma NGAL, blood samples will be taken at the preoperative, postoperative 6th and 24th hours. And the results will be recorded.

SUMMARY:
The aim of this study is to detect early renal dysfunction that may occur during the surgical procedure in geriatric patients who will undergo laparotomy surgery.

In elderly patients undergoing surgery, accurate estimation of organ function is often not possible. Accurate measurement of kidney function is vital to the routine care of patients. Determining kidney function status can predict the progression of kidney disease and prevent toxic drug levels in the body.The biochemical marker creatinine, found in serum and urine, is widely used in the estimation of GFR. Although glomerular filtration rate decreases with aging, creatinine also decreases in the elderly due to muscle loss. Even moderately elevated blood creatinine may be indicative of severe kidney failure. Creatinine clearance (CrCl) is the volume of blood plasma cleared of creatinine per unit time. It is a fast and cost-effective method for measuring kidney function. Creatine is a breakdown product of creatine phosphate found in skeletal muscle. Its production in the body depends on muscle mass. The CrCl ratio approximates the GFR calculation as it freely filters the glomerular creatine.

High serum creatinine levels and decreased CrCl ratio are usually indicators of abnormal kidney function.One of the markers of acute kidney injury is to look at plasma NGAL values. Plasma NGAL (neutrophil gelatinase associated lipocalin) increases in response to damaged kidney status and can predict acute kidney injury as an early marker. Data on investigating plasma NGAL values as a predictive biomarker of acute kidney injury in patients undergoing non-cardiovascular surgery are very limited NGAL is produced from the epithelium of kidneys, lungs, colon, liver, adipose tissue, and inflammatory cells. NGAL is elevated in serum and urine after acute tubular injury, making it possible to diagnose kidney damage within 2 hours of injury. However, the increase of other traditional markers such as creatinine may be delayed for up to 48 hours after acute kidney injury.To determine the roles of primary outcome serum creatinine, creatinine clearance rates and plasma NGAL levels in the diagnosis of acute renal failure

DETAILED DESCRIPTION:
This study will be performed on 60 patients aged 64 years and older who will undergo major abdominal laparotomy surgery in Marmara University Pendik E.A.H Operating Room, whose informed consent forms have been obtained from the patients. Patients with severe cardiac and respiratory distress, liver and kidney failure, and those who did not consent to the study will not be accepted into the study.

Preoperative (0.hour baseline), postoperative 24.,48. BUN, Creatinine, Lactate values in the blood of the patients at 1 hour, and for plasma NGAL, blood samples will be taken at the preoperative, postoperative 6th and 24th hours. And the results will be recorded.

No group will be formed in the study, which includes a total of 60 patients. All patients will be anesthetized by induction of anesthesia (2 mg/kg propfol/ 1-2 mcgr/kg remifentanil/ 0.6 mg/kg rocuronium), and intraoperative inhaler Desflurane + intravenous Remifentanil will be used to provide maintenance anesthesia. Patients will be given intravenous fluids of 4-8 ml/kg/hr with PVI monitoring, if necessary, without fluid restriction.

Statistically is acceptable for the area under the ROC curve to be above 0.700. It has been determined that we need a minimum of 60 people in order to show that an area with a minimum level of 0.700 is statistically significant.

the aim of our study is to detect early renal dysfunction that may occur during the surgical procedure in geriatric patients who will undergo laparotomy surgery.

In elderly patients undergoing surgery, accurate estimation of organ function is often not possible. Accurate measurement of kidney function is vital to the routine care of patients. Determining kidney function status can predict the progression of kidney disease and prevent toxic drug levels in the body. Glomerular filtration rate measurement includes the injection of inulin and its clearance by the kidneys. However, the use of inulin is invasive, time consuming and an expensive procedure. Alternatively, the biochemical marker creatinine, found in serum and urine, is widely used in the estimation of GFR. Although glomerular filtration rate decreases with aging, creatinine also decreases in the elderly due to muscle loss. Even moderately elevated blood creatinine may be indicative of severe kidney failure. Creatinine clearance (CrCl) is the volume of blood plasma cleared of creatinine per unit time. It is a fast and cost-effective method for measuring kidney function. Creatine is a breakdown product of creatine phosphate found in skeletal muscle. Its production in the body depends on muscle mass. The CrCl ratio approximates the GFR calculation as it freely filters the glomerular creatinine. However, it is also secreted by the peritubular capillaries, causing CrCl to overestimate GFR by about 10% to 20%. Despite the marginal error, it was an accepted method for measuring GFR due to the ease of measurement of CrCl. Creatinine clearance can be estimated using serum creatinine levels. The Cockcroft-Gault (C-G) formula uses the patient's weight (kg) and gender to estimate CrCl (mg/dL). To correct for lower CrCl in females, the resulting CrCl is multiplied by 0.85 if the patient is female. The C-G formula is age dependent as the main predictor for CrCl.

eCCr = (140 - age) x (kg) x [0.85 if female] / 72 x [Serum creatinine (mg/dL)] High serum creatinine levels and decreased CrCl ratio are usually indicators of abnormal kidney function.

One of the markers of acute kidney injury is to look at plasma NGAL values. Plasma NGAL (neutrophil gelatinase associated lipocalin) increases in response to damaged kidney status and can predict acute kidney injury as an early marker. Data on investigating plasma NGAL values as a predictive biomarker of acute kidney injury in patients undergoing non-cardiovascular surgery are very limited NGAL is produced from the epithelium of kidneys, lungs, colon, liver, adipose tissue, and inflammatory cells. NGAL is elevated in serum and urine after acute tubular injury, making it possible to diagnose kidney damage within 2 hours of injury. However, the increase of other traditional markers such as creatinine may be delayed for up to 48 hours after acute kidney injury.

To determine the roles of primary outcome serum creatinine, creatinine clearance rates and plasma NGAL levels in the diagnosis of acute renal failure

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 64 years and older (ASA I-II-III class), who were to undergo major abdominal laparotomy surgery, whose consent forms were obtained, were included in the study.

Exclusion Criteria:

* Patients with severe cardiac and respiratory distress, liver and kidney failure, and those who did not consent to the study will not be accepted into the study.

Ages: 64 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
the roles of plasma NGAL levels in acute renal failure. | first 24 hours after surgery
  roles of plasma NGAL levels in the diagnosis of acute renal failure.

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

REFERENCES:
- [Derived] Orhon Ergun M, Zengin SU, Mustafayeva A, Umuroglu T. Neutrophil gelatinase associated lipocalin in predicting postoperative acute kidney injury in elderly. Ir J Med Sci. 2022 Jun;191(3):1297-1303. doi: 10.1007/s11845-021-02865-z. Epub 2021 Nov 25. PMID 34822023